CLINICAL TRIAL: NCT02837094
Title: Enhanced Epidermal Antigen Specific Immunotherapy Trial -1 (EE-ASI-1): A Phase 1a Study of Gold Nanoparticles Administered Intradermally by Microneedles to Deliver Immunotherapy With a Proinsulin Derived Peptide in Type 1 Diabetes
Brief Title: Enhanced Epidermal Antigen Specific Immunotherapy Trial -1
Acronym: EE-ASI-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SPON1455-15
Record Dates: First submitted 2016-07-04; First posted 2016-07-19 (Estimated); Last update posted 2023-03-31 (Actual); Status verified 2021-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Safety of C19A3 GNP (general safety and induction of hypersensitivity). (Experimental): To assess general safety different parameters were taken into account: A physical examination at screening and 0, 4, 8 and 14 weeks, a review of AEs at all visits and blood tests at screening, weeks 4, 9, 14 & 20 for full blood count; urea, electrolytes and creatinine; liver function tests; (prothrombin time, total bilirubin, total protein, albumin, AST (SGOT), SGPT (ALT), alkaline phosphatase; thyroid stimulating hormone; immunoglobulins (G, A, M); calcium; magnesium, phosphate, lipid profile (total cholesterol, LDL, HDL, triglyceride), urinalysis for pH blood, protein, urine beta-2-microglobulin and albumin/creatinine ratio at screening and visits 1, 2, 4, 5 and 6 and urine for cystatin-c was tested at visits 1, 4, 5 & 6, a urine pregnancy test in females only, at all trial visits. Subjects were observed for systemic hypersensitivity to C19-A3 GNP during the immediate period after peptide injection.
  Interventions: Drug: C19-A3 GNP

INTERVENTIONS:
Drug: C19-A3 GNP — C19A3 GNP intradermal microinjectable solution of human C19A3 proinsulin peptide coupled to gold.
  Other Names: Human C19A3 proinsulin peptide coupled to gold.

SUMMARY:
The study is a two centre, open-label, uncontrolled single group phase 1A study of C19-A3 GNP peptide (10 μg peptide equivalent content) administered via Nanopass microneedles every 28 days for 8 weeks (3 doses), with follow-up for 6 weeks (14 weeks in total from first dose). Treatment will be given into the arm at a volume of 50ul.

No blinding or randomisation will be performed. In keeping with standard phase 1 study designs, no placebo or control group is included as the primary aim is to establish whether there are any major unexpected safety issues in the use of this IMP for the first time in man. 8 subjects will be recruited at 2 centres: Cardiff, UK and Linköping, Sweden.

DETAILED DESCRIPTION:
Type 1 Diabetes is caused by the body's own white blood cells damaging the insulin producing cells in the pancreas.

The aim is to develop a treatment that can slow or stop this process by switching off the white blood cells causing the damage. The aim of this study is to investigate whether giving such a treatment involving a peptide fragment related to insulin attached to gold nanoparticles is safe with no significant side-effects.

Participants need to be:

1. Diagnosed with type 1 diabetes for more than 3 months.
2. Aged between 18 and 40 years.
3. Prescribed insulin within 1 month of diagnosis. Participants will have a blood test to assess whether they have the right tissue type for the study. If suitable, they will be asked to attend their local research centre for a general examination and further blood and urine tests. If the participant still has some insulin response after the post meal urine test they will proceed to the first injection.

Each participant will have 3 injections of the same treatment, these are given 4 weeks apart. During the treatment, participants will undergo various monitoring including blood & urine tests, mixed meal tolerance tests, lymph node biopsies. A follow up appointment will take place 6 weeks after the last injection. Possible side effects include bruising and discomfort at the site of the blood test and lymph node tests, local redness and swelling reactions at the site of the injections, severe allergic reaction to the injection requiring treatment, such as steroids, adrenaline or fluids.

Participants will have more time with staff members to discuss their diabetes and ask questions than at a routine clinic appointment. It is not known whether receiving the gold particle-peptide injections will be of benefit, as this is the first study where the treatment is being used in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes for > 3 months (dated from the first insulin injection).
2. Commenced on insulin treatment within 1 month of diagnosis.
3. Age 16 to 40 years
4. 2 hour post-meal UCPCR > 0.53 nmol/mmol on at least one occasion (maximum 3 tests on different days)
5. Possession of 0401 allele at the HLA-DRB1 gene locus
6. The following birth control methods should be used (considered highly effective with a failure rate of less than 1% per year when used consistently and correctly]:

   * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

     * oral
     * intravaginal
     * transdermal
   * progestogen-only hormonal contraception associated with inhibition of ovulation:

     * oral
     * injectable
     * implantable
   * intrauterine device (IUD)
   * intrauterine hormone-releasing system (IUS)
   * bilateral tubal occlusion
   * vasectomised partner (provided that the partner is the sole sexual partner of the trial participant and that medical assessment of azoospermia has been confirmed)
   * Sexual abstinence (defined as refraining from hetrosexual intercourse during the duration of the trial)
7. Written and witnessed informed consent to participate.

Exclusion criteria

1. HbA1c > 86mmol/L (10%).
2. Females who are pregnant, breast-feeding or not using adequate forms of contraception.
3. Previous diagnosis of renal disease including glomerulonephritis or nephropathy.
4. Raised serum creatinine or abnormal urine albumin/creatinine ratio (ACR) (values above the laboratory reference range). If the initial ACR is raised, this should be repeated on two further occasions as first morning samples. The subject can be included if both of these samples are negative (within the reference range).
5. Use of immunosuppressive or immunomodulatory therapies, including systemic steroids within 1 month prior to receiving the IMP and any monoclonal antibody therapy given for any indication. Note that previous exposure to proinsulin peptide C19-A3 in a clinical trial is an exclusion criterion.
6. Use of cannabis within one month prior to trial entry.
7. Use of any hypoglycaemia agents other than insulin, for more than 6 weeks, at any time prior to trial entry.
8. Use of inhaled insulin.
9. Known alcohol abuse, drug abuse, HIV or hepatitis.
10. Allergies to drug components or any excipients.
11. Any other medical condition which, in the opinion of investigators, could affect the safety of the subject's participation or outcomes of the study, including immunocompromised states and autoimmune conditions.
12. Subjects should not have had immunisations (flu and others) for 1 month prior to trial entry and should not receive any during their time in the trial
13. Recent subject's involvement in other research studies which, in the opinion of investigators, may adversely affect the safety of the subjects or the results of the study.
14. Abnormal ECG findings.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
To examine the risk of C19A3 GNP administration in terms of general safety and induction of hypersensitivity. | 4 months
  A physical examination will be conducted at screening and 0, 4, 8 and 14 weeks. A review of AEs will be performed at all visits and blood will be drawn at screening, weeks 4, 9, 14 & 20 to examine the full blood count; urea, electrolytes and creatinine; liver function tests; (prothrombin time, total bilirubin, total protein, albumin, AST (SGOT), SGPT (ALT), alkaline phosphatase; thyroid stimulating hormone; immunoglobulins (G, A, M); calcium; magnesium, phosphate, lipid profile (total cholesterol, LDL, HDL, triglyceride). Urinalysis for pH blood, protein, urine beta-2-microglobulin and albumin/creatinine ratio will be done at screening and visits 1, 2, 4, 5 and 6 and urine for cystatin-c will be collected at visits 1, 4, 5 & 6. A urine pregnancy test will be completed in females only, at all trial visits. Induction of hypersensitivity to C19-A3 GNP will be assessed by a period of observation of subjects and during the immediate period after peptide injection.

SECONDARY OUTCOMES:
To study the feasibility of delivering C19A3 GNP via microneedles to humans. | 4 months
  By using the ultra short needles the antigen can be delivered into the superficial layers of the skin reliably with direct (perpendicular) injection. This approach has the advantage that it ensures intradermal rather than subcutaneous delivery ensuring high efficiency. At visits 1, 1b, 3b, 4, 5 and 6 blood and urine samples will be taken for gold concentrations to enable assessment of gold excretion.
To study the immune responses to C19A3 GNP generated in blood. | 4 months
  Measured as follows:
  T cell responses to C19-A3 GNP as determined by changes from baseline of interferon gamma following treatment.
To study the immune responses to C19A3 GNP generated in the draining (axillary) lymph node. | 4 months
  Measured as follows:
  T cell responses to C19-A3 GNP as determined by changes from baseline of interferon gamma in draining axillary lymph node before treatment and following the last treatment administration.

CONTACTS AND LOCATIONS:
Overall Officials: Colin M Dayan, MA FRCP PhD, Study Director — Cardiff University
Locations (1):
- Cardiff and Vale University Health Board, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tatovic D, McAteer MA, Barry J, Barrientos A, Rodriguez Terradillos K, Perera I, Kochba E, Levin Y, Dul M, Coulman SA, Birchall JC, von Ruhland C, Howell A, Stenson R, Alhadj Ali M, Luzio SD, Dunseath G, Cheung WY, Holland G, May K, Ingram JR, Chowdhury MMU, Wong FS, Casas R, Dayan C, Ludvigsson J. Safety of the use of gold nanoparticles conjugated with proinsulin peptide and administered by hollow microneedles as an immunotherapy in type 1 diabetes. Immunother Adv. 2022 Jan 27;2(1):ltac002. doi: 10.1093/immadv/ltac002. eCollection 2022. PMID 35919496

DOCUMENTS (2):
  • Study Protocol (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT02837094/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT02837094/SAP_001.pdf